CLINICAL TRIAL: NCT03541694
Title: Passive Enhanced Safety Surveillance of the Live Attenuated Yellow Fever Virus Vaccine Stamaril® in Korea
Brief Title: Passive Enhanced Safety Surveillance of Stamaril® Vaccine in Korea
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: STA10
Record Dates: First submitted 2018-04-23; First posted 2018-05-30 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2018-07

CONDITIONS: Yellow Fever
Keywords: Yellow fever; Stamaril®
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Stamaril® — Routine vaccination with Stamaril yellow fever vaccine

SUMMARY:
This is a passive enhance safety surveillance (ESS) of Stamaril® vaccine in Korea. The objective is to collect suspected related adverse events following vaccination with Stamaril® in routine practice.

DETAILED DESCRIPTION:
This ESS replaces the routing post-marketing surveillance required after product approval in Korea.

ELIGIBILITY:
Vaccination with Stamaril® vaccine in routine practice in Korea

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have been vaccinated against yellow fever with Stamaril® vaccine in Korean yellow fever vaccination centers during the enhanced surveillance period.
Sampling Method: Non-Probability Sample
Enrollment: 622 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting suspected related adverse events | Within 30 days after vaccination
  Spontaneous reporting of suspected related adverse events

SECONDARY OUTCOMES:
Number of participants reporting suspected serious related adverse events | Within 30 days after vaccination
  Spontaneous reporting of serious suspected related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Sanofi Pasteur Investigational Site 001, Seoul, South Korea